CLINICAL TRIAL: NCT03240575
Title: A Randomized, Double-blind, Double-dummy, Active-controlled, Multi-center, Parallel Group Study to Show the Superiority in Lung Function of 12 Weeks Once Daily Treatment With Orally Inhaled Tiotropium+Olodaterol Fixed Dose Combination Delivered by the Respimat® Inhaler vs. 12 Weeks Twice Daily Treatment With Fluticasone Propionate+Salmeterol Fixed Dose Combination Delivered by the Diskus® in Patients With Chronic Obstructive Pulmonary Disease (COPD) [ENERGITO® 2]
Brief Title: The ENERGITO® 2 Study Compares 2 Inhaled Medicines for Chronic Obstructive Pulmonary Disease (COPD). One Medicine is a Combination of Tiotropium and Olodaterol (Stiolto®) Taken Using the Respimat® Inhaler and the Other Medicine is a Combination of Fluticasone and Salmeterol Taken Using the Diskus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1237-0063
Record Dates: First submitted 2017-07-27; First posted 2017-08-07 (Actual); Results first posted 2020-04-16 (Actual); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide; olodaterol; Fluticasone; Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tiotropium + Olodaterol fixed dose combination (Experimental)
  Interventions: Drug: Tiotropium; Drug: Olodaterol
- Fluticasone propionate + Salmeterol fixed dose combination (Active Comparator)
  Interventions: Drug: Fluticasone propionate; Drug: Salmeterol

INTERVENTIONS:
Drug: Tiotropium — Fixed Dose Combination
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO
  Arms: Tiotropium + Olodaterol fixed dose combination
Drug: Olodaterol — Fixed Dose Combination
  Other Names: INSPIOLTO, SPIOLTO, STIOLTO, VAHELVA, YANIMO
  Arms: Tiotropium + Olodaterol fixed dose combination
Drug: Fluticasone propionate — Fixed Dose Combination
  Arms: Fluticasone propionate + Salmeterol fixed dose combination
Drug: Salmeterol — Fixed Dose Combination
  Arms: Fluticasone propionate + Salmeterol fixed dose combination

SUMMARY:
The primary objective of the trial is to show superiority in lung function of once daily (2 inhalations) treatment with orally inhaled tiotropium+olodaterol fixed dose combination to twice daily (one inhalation) treatment with fluticasone propionate+salmeterol fixed dose combination over 12 weeks in patients with Chronic Obstructive Pulmonary Disease (COPD).

A Digital Health (DH) exploratory study has been integrated into the main study as a site specific study. The DH exploratory study will be performed at a single site; the site is also participating in the main study. The DH exploratory study site will enter (randomize) approximately 20 patients (subjects) (in addition to the patients to be enrolled in the main study at this site). The patients enrolled in the DH exploratory study are not considered to be part of the main study (i.e. data collected in the DH exploratory study will be analyzed separately from the data collected in the main study).

ELIGIBILITY:
Inclusion Criteria:

* All patients must sign an informed consent consistent with FDA regulations prior to participation in the trial, which includes medication washout and restrictions.
* All patients must have a diagnosis of chronic obstructive pulmonary disease and must meet the following spirometric criteria:

  -- Patients with a post-bronchodilator 30% ≤ Forced Expiratory Volume in one second (FEV1) <80% of predicted normal (European Coal and Steel Community( ECSC)); and a post-bronchodilator FEV1/Forced Vital Capacity (FVC) <70% at Visit 1
* Male or female patients, 40 years of age or older.
* Patients must be current or ex-smokers with a smoking history of more than 10 pack years. Patients who have never smoked cigarettes must be excluded.
* Patients must be able to perform, according to investigator's judgment, all trial related procedures including:

  * Technically acceptable pulmonary function tests (spirometry)
  * Completion of study questionnaires
* Patients must be able to inhale medication in a competent manner (in the opinion of the investigator) from the Respimat® and Diskus® inhalers and from a metered dose inhaler (MDI).

Exclusion Criteria:

* Patients with a significant disease other than Chronic Obstructive Pulmonary Disease (COPD); a significant disease is defined as a disease which, in the opinion of the investigator, may (i) put the patient at risk because of participation in the study, (ii) influence the results of the study, or (iii) cause concern regarding the patient's ability to participate in the study.
* Patients who have had a COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization in the last 3 months prior to Visit 1 and/or between Visit 1 and Visit 2.
* Patients with a history of asthma. For patients with allergic rhinitis or atopy, source documentation is required to verify that the patient does not have asthma. If a patient has a total blood eosinophil count ≥ 600/mm3, source documentation is required to verify that the increased eosinophil count is related to a nonasthmatic condition.

Patients with any of the following conditions:

* A diagnosis of thyrotoxicosis (due to the known class side effect profile of ß2-agonists).
* A diagnosis of paroxysmal tachycardia (>100 beats per minute) (due to the known class side effect profile of ß2-agonists).
* A history of myocardial infarction within 1 year of screening visit (Visit 1).
* Unstable or life-threatening cardiac arrhythmia.
* Hospitalization for heart failure within the past year.
* Known active tuberculosis.
* A malignancy for which patient has undergone resection, radiation therapy or chemotherapy within last five years (patients with treated basal cell carcinoma are allowed).
* A history of life-threatening pulmonary obstruction.
* A history of cystic fibrosis.
* Clinically evident bronchiectasis.
* A history of significant alcohol or drug abuse.
* Patients who have undergone thoracotomy with pulmonary resection (patients with a history of thoracotomy for other reasons should be evaluated as per the first exclusion criterion).
* Patients being treated with oral or patch β-adrenergics.
* Patients being treated with oral corticosteroid medication within 6 weeks prior to Visit 1.
* Patients who regularly use daytime oxygen therapy for more than one hour per day and in the investigator's opinion will be unable to abstain from the use of oxygen therapy during clinic visits.
* Patients who have completed a pulmonary rehabilitation program in the six weeks prior to the screening visit (Visit 1) or patients who are currently in a pulmonary rehabilitation program.
* Patients who have taken an investigational drug within one month, six half-lives or within the wash out period (whichever is greater) prior to screening visit (Visit 1).
* Patients with known hypersensitivity to β-adrenergic drugs, BAC, EDTA, or any other component of the Respimat® inhalation solution. In addition, patients with known hypersensitivity to Lactose monohydrate (which contains milk proteins).
* Pregnant or nursing women.
* Women of childbearing potential not using a method of birth control classified at least as "acceptable". Female patients will be considered to be of childbearing potential unless surgically sterilized by hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or post-menopausal (defined as no menses for 12 months without an alternative medical cause). Tubal ligation is NOT a method of permanent sterilisation.
* Patients who have previously been randomized in this study or are currently participating in another study.
* Patients who are unable to comply with pulmonary medication restrictions prior to randomization.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2017-08-14 (Actual); Primary Completion 2019-04-08 (Actual); Study Completion 2019-05-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Jasper Summit Research, LLC, Jasper, Alabama
  - Clinical Trial Connection, Flagstaff, Arizona
  - California Research Medical Group, Inc., Fullerton, California
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - California Medical Research Associates Inc., Northridge, California
  - IMMUNOe Research Centers, Centennial, Colorado
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Bioclinica Research, Orlando, Florida
  - IMIC, Inc, Palmetto Bay, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Duluth Biomedical Research, Duluth, Georgia
  - DC Pulmonary Medicine, Marietta, Georgia
  - New Orleans Center for Clinical Research, New Orleans, Louisiana
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Pulmonary Rsrch Inst of SE MI, Farmington Hills, Michigan
  - Minnesota Lung Center and Sleep Institute, Edina, Minnesota
  - Clinical Research Institute Inc, Minneapolis, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Northwell Health, New Hyde Park, New York
  - Gastonia Pharmaceutical Research, LLC, Gastonia, North Carolina
  - Hendersonville Pharmaceutical Research, Hendersonville, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Bernstein Clinical Rsrch Ctr, Cincinnati, Ohio
  - Aventiv Research Inc., Columbus, Ohio
  - Aventiv Research Inc., Dublin, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - IPS Research Company, Oklahoma City, Oklahoma
  - Arcuri Clinical Research, LLC, Philadelphia, Pennsylvania
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
  - VitaLink Research - Easley, Easley, South Carolina
  - VitaLink Research -Gaffney, Gaffney, South Carolina
  - VitaLink Research, Greenville, South Carolina
  - Vita Link Research- Rock Hill, Rock Hill, South Carolina
  - South Carolina Pharma Rsrch, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - Centex Studies, Inc., Houston, Texas
  - Advanced Clinical Research Associates, Plano, Texas
  - Sherman Clinical Research, Sherman, Texas
  - DM Clinical Research, Tomball, Texas
  - Pulmonary Associates of Richmond, Inc., Richmond, Virginia
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - Morgantown Pulmonary ClinRsrch, Morgantown, West Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study compares treatment tiotropium+olodaterol (5μg/5μg) once daily FDC to Fluticasone propionate+Salmeterol (250μg/50μg) twice daily FDC over 12 weeks in patients with COPD. A Digital Health (DH)-study has been integrated a site specific study. The patients enrolled in the DH-study are not considered to be part of the main study.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and non of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- Tiotropium+Olodaterol (5μg/5μg) - Main Study: 2 inhalations of fixed dose combination (FDC) of 2.5 microgram (μg) tiotropium and 2.5μg olodaterol (T+O) (total 5μg/5μg) were administered orally once daily in the morning via RESPIMAT inhaler over a treatment period of 12 weeks in patients with Chronic Obstructive Pulmonary Disease (COPD). Patients enrolled in the main study were not eligible to participate in the DH study.
- Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study: 2 inhalations of fixed dose combination (FDC) of 250μg fluticasone propionate and 50μg salmeterol (F+S) (total 500μg/100μg) were administered orally twice daily in the morning and in the evening (12h after morning dose) via Diskus inhaler over a treatment period of 12 weeks in patients with Chronic Obstructive Pulmonary Disease (COPD). Patients enrolled in the main study were not eligible to participate in the DH study.
- Tiotropium+Olodaterol (5μg/5μg) - DH-study: 2 inhalations of fixed dose combination (FDC) of 2.5 microgram (μg) tiotropium and 2.5μg olodaterol (T+O) (total 5μg/5μg) were administered orally once daily in the morning via RESPIMAT inhaler over a treatment period of 12 weeks in patients with Chronic Obstructive Pulmonary Disease (COPD). Patients enrolled in the DH study were not eligible to participate in the main study.
- Fluticasone Propionate+Salmeterol (500μg/100μg) - DH-study: 2 inhalations of fixed dose combination (FDC) of 250μg fluticasone propionate and 50μg salmeterol (F+S) (total 500μg/100μg) were administered orally twice daily in the morning and in the evening (12h after morning dose) via Diskus inhaler over a treatment period of 12 weeks in patients with Chronic Obstructive Pulmonary Disease (COPD). Patients enrolled in the DH study were not eligible to participate in the main study.
Period: Overall Study
Arm/Group | Tiotropium+Olodaterol (5μg/5μg) - Main Study | Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study | Tiotropium+Olodaterol (5μg/5μg) - DH-study | Fluticasone Propionate+Salmeterol (500μg/100μg) - DH-study
Started | 146 | 145 | 6 | 5
Completed | 144 | 131 | 6 | 3
Not Completed | 2 | 14 | 0 | 2
Not completed — Adverse Event | 0 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 11 | 0 | 1
Not completed — Other | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): All randomized patients who had taken at least one dose of study drug were included in the treated set.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tiotropium+Olodaterol (5μg/5μg) - Main Study | Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study | Tiotropium+Olodaterol (5μg/5μg) - DH-study | Fluticasone Propionate+Salmeterol (500μg/100μg) - DH-study | Total
Number analyzed (Participants) | 146 | 145 | 6 | 5 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.95 (8.32) | 64.74 (7.33) | 71.00 (4.77) | 60.00 (4.58) | 63.44 (7.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 62 | 1 | 4 | 139
  Male | 74 | 83 | 5 | 1 | 163
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 0 | 0 | 4
  Not Hispanic or Latino | 144 | 143 | 6 | 5 | 298
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 14 | 16 | 0 | 0 | 30
  White | 132 | 127 | 6 | 5 | 270
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve From 0 to 24 Hours (AUC0-24) Response (Change From Baseline) [L] After 12 Weeks of Treatment
Description: Forced Expiratory Volume in one second (FEV1) Area under the Curve from 0 to 24 hours (AUC0-24) response (change from baseline) [L] after 12 weeks of treatment. FEV1 AUC0-24 was calculated as the area under the FEV1-time curve from 0-24 hours post-dose using the trapezoidal rule, divided by the duration (24 hours) and reported in liters. FEV1 AUC0-24 response (change from baseline) was defined as FEV1 AUC0-24 mius baseline FEV1.
Time Frame: 1 hours (h) and 10 minutes (min) before first dose at day1 of weeks 1 for baseline.10 min before and 30 min, 1 h, 2h, 3h, 4h, 6h, 8h, 10h, 11h 50min, 12h 30 min, 13h, 14h, 22h, 23h, and 24h post morning dose at week 12.
Population: Full Analysis Set (FAS): FAS included all patients in the TS who had baseline and at least one post-baseline measurement for at least one efficacy parameter. The Mixed-effects model repeated measurement (MMRM) model defined the participants who contributed to the model.
Measure: Mean (Standard Error); unit: Litre*hours (L*h)
Arm/Group | Tiotropium+Olodaterol (5μg/5μg) - Main Study | Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study | Tiotropium+Olodaterol (5μg/5μg) - DH-study | Fluticasone Propionate+Salmeterol (500μg/100μg) - DH-study
Number analyzed (Participants) | 145 | 138 | 6 | 4
Litre*hours (L*h) | 0.174 (0.019) | 0.122 (0.019) | NA (NA) — Due to the small number of subjects and due to the many out of window test assessments, the primary endpoint could not be evaluated. | NA (NA) — Due to the small number of subjects and due to the many out of window test assessments, the primary endpoint could not be evaluated.
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (5μg/5μg) - Main Study vs Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study; Test type: Superiority; p = 0.0543, Mixed-effects model repeated measures; Treatment, visit and treatment by visit interaction as fixed effects, and baseline as well as baseline by visit interaction as covariates; Mean Difference (Net) = 0.052, 95% CI 2-sided [-0.001 to 0.105], Standard Error of Mean 0.027

2. Secondary Outcome: Forced Expiratory Volume in One Second (FEV1) Area Under the Curve From 0 to 12 Hours (AUC0-12) Response (Change From Baseline) [L] After 12 Weeks of Treatment
Description: Forced Expiratory Volume in one second (FEV1) Area under the Curve from 0 to 12 hours (AUC0-12) response (change from baseline) [L] after 12 weeks of treatment.
  FEV1 AUC0-12 was calculated as the area under the FEV1-time curve from 0-12 hours post-dose using the trapezoidal rule, divided by the duration (12 hours) and reported in liters. FEV1 AUC0-12 response (change from baseline) was defined as FEV1 AUC0-12 minus baseline FEV1.
Time Frame: 1 hours (h) and 10 minutes (min) before first dose at day1 of weeks 1 for baseline. 10 min before and 30 min, 1 h, 2h, 3h, 4h, 6h, 8h, 10h, 11h 50min post morning dose at week 12.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre*hours (L*h)
Arm/Group | Tiotropium+Olodaterol (5μg/5μg) - Main Study | Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study | Tiotropium+Olodaterol (5μg/5μg) - DH-study | Fluticasone Propionate+Salmeterol (500μg/100μg) - DH-study
Number analyzed (Participants) | 145 | 138 | 6 | 3
Litre*hours (L*h) | 0.237 (0.019) | 0.147 (0.020) | NA (NA) — Based on the exploratory study design of the DH-study and the small number of patients, Endpoints were planned to be analyzed descriptively. | NA (NA) — Based on the exploratory study design of the DH-study and the small number of patients, Endpoints were planned to be analyzed descriptively.
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (5μg/5μg) - Main Study vs Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study; Test type: Superiority; p = 0.0011, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.090, 95% CI 2-sided [0.037 to 0.144], Standard Error of Mean 0.027

3. Secondary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) Response (Change From Baseline) [L] After 12 Weeks Treatment
Description: Trough Forced Expiratory Volume in one second (FEV1) response (change from baseline) [L] after 12 weeks treatment. Trough FEV1 was defined as the mean of the FEV1 value measured at 23 hours and at 24 hours after the trial medication administration. Through FEV1 response (change from baseline) was defined as trough FEV1 minus baseline FEV1.
Time Frame: At 23 h and 24 h post dose at baseline and at 23h and 24 h post dose at week 12.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium+Olodaterol (5μg/5μg) - Main Study | Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study | Tiotropium+Olodaterol (5μg/5μg) - DH-study | Fluticasone Propionate+Salmeterol (500μg/100μg) - DH-study
Number analyzed (Participants) | 145 | 138 | 6 | 3
Litre (L) | 0.118 (0.019) | 0.114 (0.019) | NA (NA) — Based on the exploratory study design of the DH-study and the small number of patients, Endpoints were planned to be analyzed descriptively. | NA (NA) — Based on the exploratory study design of the DH-study and the small number of patients, Endpoints were planned to be analyzed descriptively.
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (5μg/5μg) - Main Study vs Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study; Test type: Superiority; p = 0.8593, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.005, 95% CI 2-sided [-0.048 to 0.058], Standard Error of Mean 0.027

4. Secondary Outcome: Peak 0-3 Hours Forced Expiratory Volume in One Second (FEV1) Response (Change From Baseline) [L] After 12 Weeks Treatment
Description: Peak 0-3 hours Forced Expiratory Volume in one second (FEV1) response (change from baseline) [L] after 12 weeks treatment. Peak 0-3h was defined as the maximum value measured within the first three hours post doing.
Time Frame: 30 minutes, 1 h, 2h and 3h post dose at baseline and week 12.
Population: as for outcome 1
Measure: Mean (Standard Error); unit: Litre (L)
Arm/Group | Tiotropium+Olodaterol (5μg/5μg) - Main Study | Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study | Tiotropium+Olodaterol (5μg/5μg) - DH-study | Fluticasone Propionate+Salmeterol (500μg/100μg) - DH-study
Number analyzed (Participants) | 144 | 138 | 6 | 3
Litre (L) | 0.341 (0.021) | 0.243 (0.021) | NA (NA) — Based on the exploratory study design of the DH-study and the small number of patients, Endpoints were planned to be analyzed descriptively. | NA (NA) — Based on the exploratory study design of the DH-study and the small number of patients, Endpoints were planned to be analyzed descriptively.
Statistical Analysis 1: Comparison: Tiotropium+Olodaterol (5μg/5μg) - Main Study vs Fluticasone Propionate+Salmeterol (500μg/100μg) - Main Study; Test type: Superiority; p = 0.0010, Mixed-effects model repeated measures; [statistical method as in outcome 1, analysis 1]; Mean Difference (Net) = 0.098, 95% CI 2-sided [0.040 to 0.156], Standard Error of Mean 0.029

ADVERSE EVENTS:
Time Frame: From screening visit (28 days before treatment start) until end of follow up period (up to 105 days).
Description: Safety analysis is reported for TS of both studies. Participants of each particular treatment arm in main and DH-study were combined in one particular treatment arm for adverse event reporting.
Groups:
- Tiotropium+Olodaterol (5μg/5μg): Once daily treatment of orally inhaled tiotropium + olodaterol (T+O) (5μg/5μg) fixed dose combination (FDC) over 12 weeks in patients with Chronic Obstructive Pulmonary Disease (COPD). Patients from Main and DH-study combined.
- Fluticasone Propionate+Salmeterol (500μg/100μg): Twice daily treatment of orally inhaled fluticasone propionate + salmeterol (F+S) (250μg/50μg) fixed dose combination (FDC) over 12 weeks in patients with Chronic Obstructive Pulmonary Disease (COPD). Patients from Main and DH-study combined.
Arm/Group | Tiotropium+Olodaterol (5μg/5μg) | Fluticasone Propionate+Salmeterol (500μg/100μg)
All-Cause Mortality (participants affected / at risk) | 0/152 | 0/150
Serious Adverse Events (participants affected / at risk) | 6/152 | 3/150
Other Adverse Events (participants affected / at risk) | 8/152 | 15/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium+Olodaterol (5μg/5μg) (N=152) | Fluticasone Propionate+Salmeterol (500μg/100μg) (N=150)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc compression (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the oral cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tiotropium+Olodaterol (5μg/5μg) (N=152) | Fluticasone Propionate+Salmeterol (500μg/100μg) (N=150)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 8 | 15

LIMITATIONS AND CAVEATS:
The objectives of the DH-study were exploratory. The DH-study aimed to gather information and experience about the feasibility of a remote trial in this indication, and was not designed to support treatment comparisons.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT03240575/SAP_000.pdf
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/75/NCT03240575/Prot_001.pdf